CLINICAL TRIAL: NCT03917719
Title: An Open-Label Extension Study of Edasalonexent in Pediatric Patients With Duchenne Muscular Dystrophy
Brief Title: An Open-Label Extension Study of Edasalonexent in Boys With Duchenne Muscular Dystrophy
Acronym: GalaxyDMD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Phase 3 PolarisDMD trial did not meet the primary endpoint. As a result, activities related to the development of edasalonexent have stopped including the CAT-1004-302 Open-Label Study of Edasalonexent in Boys With Duchenne Muscular Dystrophy
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-1004-302
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases; DMD; dystrophin; dystrophy; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases | interventions — edasalonexent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose 1 (Experimental): Edasalonexent 100mg/kg/day. Capsules taken by mouth three times per day.
  Interventions: Drug: Edasalonexent

INTERVENTIONS:
Drug: Edasalonexent — 100 mg/kg/day
  Other Names: Edasa; CAT-1004

SUMMARY:
The GalaxyDMD study is a global Phase 3, open-label, treatment extension study to evaluate the safety, tolerability, and durability of effect in long-term dosing of edasalonexent in pediatric patients with a genetically confirmed diagnosis of DMD. Patients who completed CAT-1004-201 or CAT-1004-301 or siblings of these boys from 4-12 years of age (up to 13th birthday) will be enrolled.

Edasalonexent is an orally administered small molecule that inhibits NF-kB, which is a key link between loss of dystrophin and disease pathology and plays a fundamental role in the initiation and progression of skeletal and cardiac muscle disease in DMD.

DETAILED DESCRIPTION:
The study includes a 104-week open-label treatment period with edasalonexent. Patients who completed CAT-1004-201 or CAT-1004-301 and eligible siblings of these boys will be enrolled in this trial.

ELIGIBILITY:
For Patients who Completed CAT-1004-201 or CAT-1004-301:

Inclusion Criteria:

* Written consent/assent by patient and/or legal guardian as per regional and/or Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements
* Completion of either CAT-1004-201 or CAT-1004-301

Exclusion Criteria:

* In the Investigator's opinion, unwilling or unable for any reason to complete all study assessments and laboratory tests and comply with scheduled visits, administration of drug, and all other study procedures

For Siblings of Patients who Completed CAT-1004-201 or CAT-1004-301:

Inclusion Criteria:

* Written consent/assent by patient and/or legal guardian as per regional and/or Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements
* A sibling of a patient who completed either CAT-1004-201 or CAT-1004-301
* Diagnosis of DMD based on a clinical phenotype with increased serum creatine kinase (CK) and documentation of mutation(s) in the dystrophin gene known to be associated with a DMD phenotype
* Followed by a doctor or medical professional who coordinates Duchenne care on a regular basis and willingness to disclose patient's study participation with medical professionals

Exclusion Criteria:

* Use of oral corticosteroids at screening; use of inhaled, intranasal, and topical corticosteroids is permitted
* Use of another investigational drug, idebenone, or dystrophin-focused therapy within 4 weeks. Exception: Patients who are currently on or plan to initiate treatment with approved oligonucleotide exon-skipping therapies, and expected to continue treatment throughout the study, will be eligible
* Use of the following within 4 weeks prior to Day 1: immunosuppressive therapy, anticoagulants, cyclosporine, dihydroergotamine, ergotamine, fentanyl, alfentanil, pimozide, quinidine, sirolimus or tacrolimus
* Use of human growth hormone within 3 months prior to Day 1
* Other prior or ongoing significant medical conditions

Ages: 4 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of long-term treatment with edasalonexent measured by number of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 104 Weeks

SECONDARY OUTCOMES:
Durability of effects of edasalonexent on physical function as measured by the North Star Ambulatory Assessment (NSAA) | 104 Weeks
Durability of effects of edasalonexent on physical function as measured by the 10-meter walk/run test | 104 Weeks
Durability of effects of edasalonexent on physical function as measured by the time to stand from supine | 104 Weeks
Durability of effects of edasalonexent on physical function as measured by the 4-stair climb | 104 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Donovan, MD, PhD, Study Chair — Catabasis Pharmaceuticals
Locations (23):
- United States (15):
  - UC Davis, Sacramento, California
  - Rare Disease Research, LLC, Atlanta, Georgia
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Las Vegas Clinic, Las Vegas, Nevada
  - Shriners Hospital for Children, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Royal Children's Hospital, Parkville, Victoria, Australia
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada
- Germany (2):
  - University of Hamburg, Hamburg
  - University of Munich, Munich
- Queen Silvia Children's Hospital, Gothenburg, Sweden
- United Kingdom (3):
  - Bristol Children's Hospital, Bristol
  - Great Ormond Street Hospital (GOSH), London
  - Royal Manchester Children's Hospital, Manchester